CLINICAL TRIAL: NCT01604564
Title: KOPOF Registry (Patients Characteristics, Operative Data, Postoperative Outcome, Functional Postoperative Recovery ) of Patients in Which a Pouch Has Been Created Due to Colitis Ulcerosa (CU) or Familial Adenomatous Polyposis(FAP)
Brief Title: Registry With Information About Colitis Ulcerosa and Familial Adenomatous Polyposis Patients
Acronym: KOPOF
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S-54228
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Colitis,Ulcerative; Adenomatous Polyposis Coli; Reservoir, Ileoanal
Keywords: Registry; Colitis Ulcerosa (CU); Familial Adenomatous Polyposis(FAP); IPAA
MeSH Terms: conditions — Colitis, Ulcerative; Adenomatous Polyposis Coli

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Colitis Ulcerosa: Colitis Ulcerosa With creation of IPAA
- Familial Adenomatous Polyposis: Familial Adenomatous Polyposis with creation of IPAA

SUMMARY:
The purpose of this registry is to collect information about patients in which a pouch has been created to improve in the future the quality of the surgery of the pouch.

DETAILED DESCRIPTION:
To improve the quality of the surgery of the pouch created in CU and FAP patients, the following information will be collected: Patients Characteristics, Operative Data, Postoperative Outcome and Functional Postoperative Recovery.

ELIGIBILITY:
Inclusion Criteria:

* Colitis Ulcerosa or Familial Adenomatous Polyposis Patients With IPAA

Exclusion Criteria:

* No

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Colitis Ulcerosa or Familial Adenomatous Polyposis Patients who have undergone a restorative proctocolectomy with creation of an ileoanal pouche
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2012-05; Primary Completion 2018-07 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of postoperatieve recovery | 1 YEAR
  STANDARD QUESTIONS AT 1, 3, 6 AND 12 MONTHS FU

CONTACTS AND LOCATIONS:
Overall Officials: André JL D'Hoore, PhD, Principal Investigator — University Clinics Gasthuisberg Department of Abdominal Surgery
Locations (1):
- University Clinics Gasthuisberg, Leuven, Flemish Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No